CLINICAL TRIAL: NCT05748041
Title: Multiparametric Approach to Identify a CMR-based Tricuspid Regurgitation Classification
Acronym: TRAC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Giulia Pasqualin, Investigator, IRCCS Policlinico S. Donato
Other Study IDs: TRAC
Record Dates: First submitted 2023-02-01; First posted 2023-02-28 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Tricuspid Regurgitation Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aims of this study are:

1. to explore a novel 2D-Cardiovascular magnetic resonance (CMR) indirect method for tricuspid regurgitation (TR) quantification (ATRIAL method) relying on right atrium variables, and assess its agreement with the traditional indirect method (involving right ventricle variables) and the direct method (based on through-plane phase contrast (PC) sequences on the tricuspid valve);
2. to assess the agreement of TR volume (RVol) and regurgitant fraction quantification from 2D-CMR methods with transthoracic echocardiography and 4DF-CMR methods;
3. to assess the diagnostic performance of 2D-CMR in classifying TR, in terms of RVol and regurgitant fraction, with respect to echocardiographic transthoracic echocardiography grades.

ELIGIBILITY:
Inclusion Criteria:

* patients aged ≥ 18 years with the diagnosis of al least mild-degree tricuspid regurgitation, who:
* patients that are scheduled for a Cardiovascular Magnetic Resonance examination in our Institution

Exclusion Criteria:

* Patients with previous surgical or transcatheter interventions on the tricuspid valve
* Patients with Ebstein's disease
* Subjects with pace-maker or intracardiac defibrillator
* Subjects with intrabody ferromagnetic material precluding patient's safety
* Patients with claustrophobia or breath-holding precluding an adequate CMR images quality
* Pregnant women

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of tricuspid regurgitation.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Estimated)
Dates: Start 2021-02-16 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
2D-CMR (different methods) | 3 years

SECONDARY OUTCOMES:
RVol and RF | 3 years

OTHER OUTCOMES:
TTE, performed within 30 days from the CMR examination | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Policlinico San Donato, San Donato Milanese, Milano, Italy